CLINICAL TRIAL: NCT07148869
Title: The Effect of Laughter Yoga Practice on Anxiety, Sleep Quality, Treatment Compliance and Satisfaction in Hypertension Patients
Brief Title: The Effect of Laughter Yoga Practice in Hypertension Patients
Acronym: HT-Laughter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kilis 7 Aralik University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, GÜLSEN KARATAŞ, Lecturer, Kilis 7 Aralik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HASAN KALYONCU UNIVERSITY
Record Dates: First submitted 2025-07-18; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Laughter Yoga
Keywords: Hypertension; Sleep Quality; laughter yoga; anxiety; treatment compliance
MeSH Terms: conditions — Hypertension; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Patient Compliance | interventions — Laughter Therapy; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: 2 group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laughter yoga group (Experimental): Patients will be divided into groups of at least 5 people according to the sample size. Laughter yoga sessions will be conducted under the leadership of the researcher in a suitable room / hall determined within the hospital. A total of 8 sessions will be applied, 2 sessions per week for 4 weeks, with each session lasting an average of 40 minutes.
  Interventions: Behavioral: LAUGHTER YOGA
- CONTROL GROUP (Placebo Comparator): there will be no application to this group
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: LAUGHTER YOGA — Patients will be divided into groups of at least 5 people according to the sample size. Laughter yoga sessions will be conducted under the leadership of the researcher in a suitable room / hall determined within the hospital. A total of 8 sessions will be applied, 2 sessions per week for 4 weeks, with each session lasting an average of 40 minutes.
  Arms: laughter yoga group
Other: control group — there will be no application to this group
  Arms: CONTROL GROUP

SUMMARY:
Hypertension (HT), which is defined as an arterial blood pressure higher than 140/90 mmHg, is an important health problem because it causes serious complications and is commonly seen in the community.

Laughter as an expression of humour has been accepted as a good medicine for centuries. It is also one of the practices used in nursing care according to the Nursing Interventions Classification (NIC). Laughter yoga developed by Dr. Madan Kataria, an Indian medical doctor, in 1995 includes deep breathing exercises, meditation, childish games and laughter without humour. In practice, individual sessions as well as group sessions can be held. It is important to form groups of at least 5 people in terms of the dynamics of the group. The first stage in laughter yoga is warm-up exercises. Hands are clapped parallel to each other, acupuncture points are stimulated by stimulating the fingertips and palms as clapping is performed, and a vocal rhythm in the form of ho, ho, ha-ha-ha is added to the last clapping movement. In the second stage, breathing exercises, the participants raise their arms to the sky as if praying, inhale and hold their breath for 4-5 seconds after deep inspiration and exhale rhythmically and slowly. The third stage includes childish games. The last stage is the stage of laughter exercises in which unreasonable laughter is thrown by imagining situations as if they did not exist. These exercises include milkshake laughter exercises, lion laughter, hot soup laughter, hugging laughter, bird laughter, etc. It is recommended that each session should be at least 20 minutes and should be applied for at least 8 weeks. At the end of the session, individuals are provided to relax by meditation.

The aim of this thesis study;

* Developing the Laughter Yoga Satisfaction Scale and
* To investigate the effect of laughter yoga practice on anxiety, sleep quality, treatment compliance and satisfaction in hypertension patients.

Hypotheses of the study H1-1: Laughter Yoga Satisfaction Scale is a valid scale. H2-1: Laughter Yoga Satisfaction Scale is a reliable scale. H3-1: Laughter yoga reduces the anxiety level of hypertension patients. H4-1: Laughter yoga improves the sleep quality of hypertension patients. H5-1: Laughter yoga increases the level of compliance with treatment in hypertension patients.

H6-1: Hypertension patients have a high level of satisfaction with laughter yoga.

H7-1: Laughter yoga has positive effects on vital signs of hypertension patients.

DETAILED DESCRIPTION:
Patient Information Form: In the form developed by the researcher as a result of literature review, some sociodemographic characteristics of the patients (age, gender, educational status, marital status, social security, employment and income status, smoking and alcohol use) were included. and medical characteristics (duration of HT diagnosis, medications used, presence of hypertension in the family, other chronic diseases) will be included.

Life Findings Record Form: The researcher will measure the patient's blood pressure, oxygen saturation, pulse and respiratory rate, body temperature 10 minutes before and 10 minutes after the laughter yoga session and record them on this form.

Pittsburgh Sleep Quality Index (PSQI): The scale consists of 18 items and 7 components. The total PDQI score is the sum of the scores of these components and the total score takes a value between 0-21. A PDQI total score >5 indicates 'poor sleep quality' and a PDQI total score <5 indicates 'good sleep quality'. The Cronbach alpha reliability coefficient of the Turkish version of the scale was found to be 0.80.

State and Trait Anxiety Inventory (STAI): The scale consists of two separate forms, a 20-item State Anxiety Scale and a 20-item Trait Anxiety Scale. The total score value obtained from the scales is between 20 and 80 points. Scores close to 80 points indicate a high level of anxiety. Scale reliability according to Kuder-Richardson reliability: 0.83 to 0.87 for Trait Anxiety Scale and 0.94 to 0.96 for State Anxiety Scale. Item reliability correlations were found between 0.34 and 0.72 for the Trait Anxiety Scale and between 0.42 and 0.85 for the State Anxiety Scale. In the scale, which measures momentary (temporary) anxiety at a reliable level, participants tick the most appropriate option from the options of "not at all", "a little", "a lot" or "completely" for each statement in the state anxiety scores. Positive scores (increasing the total anxiety score) are given for items; negative scores (decreasing the total anxiety score) are given for items. During the evaluation, a score between 1 (or -1) and 4 (or -4) is given for each item according to the positive or negative feature of the item and a constant of 50 is added to the total score to be obtained. The highest score is 80 and the lowest score is 20. The higher the total anxiety score, the higher the anxiety level of the respondent.

Hill-Bone Hypertension Treatment Compliance Scale: The four-point Likert-type scale (0=never, 1=sometimes, 2=most of the time and 3=always) consists of 14 items and has three sub-dimensions including interview, medical and nutrition. The scores that can be obtained from the scale vary between 0 (perfect agreement) and 42 (incompatible). As the score obtained from the scale increases, treatment compliance decreases. While the Cronbach alpha value of the original scale was found to be 0.84, the Cronbach alpha reliability coefficient of the Turkish version was found to be 0.83.

Laughter Yoga Satisfaction Scale: In the first stage of the research, the scale developed by the researcher and the validity-reliability study will be used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hypertension in the last one year
* Those who volunteered to participate in the study
* No problem preventing communication
* No cognitive and mental problems
* Not taking anxiolytics, antidepressants or sleeping pills
* Individuals without an additional chronic disease that may affect breathing, such as heart failure or chronic obstructive pulmonary disease

Will be included in the research.

Exclusion Criteria:

* The patient wishes to leave the study voluntarily
* Less than 80% participation of the patient in the laughter yoga programme
* Failure of the patient to participate in follow-up assessments
* The patient receives additional treatments during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Life Findings Record Form | Day 1
  The researcher will measure the patient's blood pressure, oxygen saturation, pulse and respiratory rate, body temperature 10 minutes before and 10 minutes after the laughter yoga session and record them on this form.
Sleep Quality | Day 1
  Pittsburgh Sleep Quality Index (PSQI): The Turkish validity and reliability of the scale developed by Buysse et al. to evaluate sleep quality in the last month was performed by Ağargün et al. The scale consists of 18 items and 7 components. The total PDQI score is the sum of the scores of these components and the total score takes a value between 0-21. A PDQI total score >5 indicates 'poor sleep quality' and a PDQI total score <5 indicates 'good sleep quality'. The Cronbach alpha reliability coefficient of the Turkish version of the scale was found to be 0.80.
State and Trait Anxiety Inventory | Day 1
  State and Trait Anxiety Inventory (STAI): The scale developed by Spielberger et al. (1970) was adapted to Turkish culture and validity and reliability studies were conducted by Öner and Le Compte (1983). The scale consists of two separate forms, a 20-item State Anxiety Scale and a 20-item Trait Anxiety Scale. The total score value obtained from the scales is between 20 and 80 points. Scores close to 80 points indicate a high level of anxiety. Scale reliability according to Kuder-Richardson reliability: 0.83 to 0.87 for Trait Anxiety Scale and 0.94 to 0.96 for State Anxiety Scale. Item reliability correlations were found between 0.34 and 0.72 for the Trait Anxiety Scale and between 0.42 and 0.85 for the State Anxiety Scale. In the scale, which measures momentary (temporary) anxiety at a reliable level, participants tick the most appropriate option from the options of "not at all", "a little", "a lot" or "completely" for each statement in the state anxiety scores. Positive scores (incre
Hill-Bone Hypertension Treatment Compliance | Day 1
  Hill-Bone Hypertension Treatment Compliance Scale: The Turkish validity and reliability of the scale developed by Kim et al. was performed by Karademir et al. The four-point Likert-type scale (0=never, 1=sometimes, 2=most of the time and 3=always) consists of 14 items and has three sub-dimensions including interview, medical and nutrition. The scores that can be obtained from the scale vary between 0 (perfect agreement) and 42 (incompatible). As the score obtained from the scale increases, treatment compliance decreases. While the Cronbach alpha value of the original scale was found to be 0.84, the Cronbach alpha reliability coefficient of the Turkish version was found to be 0.83.
Laughter Yoga Satisfaction | Day 4
  Laughter Yoga Satisfaction Scale: In the first phase of the study, the scale developed by the researcher and the validity-reliability study will be used. On a scale ranging from a minimum of 13 to a maximum of 65, it is shown that satisfaction increases as the score increases.

SECONDARY OUTCOMES:
Sleep Quality | four weeks later
  Pittsburgh Sleep Quality Index (PSQI): The Turkish validity and reliability of the scale developed by Buysse et al. to evaluate sleep quality in the last month was performed by Ağargün et al. The scale consists of 18 items and 7 components. The total PDQI score is the sum of the scores of these components and the total score takes a value between 0-21. A PDQI total score >5 indicates 'poor sleep quality' and a PDQI total score <5 indicates 'good sleep quality'. The Cronbach alpha reliability coefficient of the Turkish version of the scale was found to be 0.80.
State and Trait Anxiety Inventory | four weeks later
  State and Trait Anxiety Inventory (STAI): The scale developed by Spielberger et al. (1970) was adapted to Turkish culture and validity and reliability studies were conducted by Öner and Le Compte (1983). The scale consists of two separate forms, a 20-item State Anxiety Scale and a 20-item Trait Anxiety Scale. The total score value obtained from the scales is between 20 and 80 points. Scores close to 80 points indicate a high level of anxiety. Scale reliability according to Kuder-Richardson reliability: 0.83 to 0.87 for Trait Anxiety Scale and 0.94 to 0.96 for State Anxiety Scale. Item reliability correlations were found between 0.34 and 0.72 for the Trait Anxiety Scale and between 0.42 and 0.85 for the State Anxiety Scale. In the scale, which measures momentary (temporary) anxiety at a reliable level, participants tick the most appropriate option from the options of "not at all", "a little", "a lot" or "completely" for each statement in the state anxiety scores. Positive scores (incre
Hill-Bone Hypertension Treatment Compliance | four weeks later
  Hill-Bone Hypertension Treatment Compliance Scale: The Turkish validity and reliability of the scale developed by Kim et al. was performed by Karademir et al. The four-point Likert-type scale (0=never, 1=sometimes, 2=most of the time and 3=always) consists of 14 items and has three sub-dimensions including interview, medical and nutrition. The scores that can be obtained from the scale vary between 0 (perfect agreement) and 42 (incompatible). As the score obtained from the scale increases, treatment compliance decreases. While the Cronbach alpha value of the original scale was found to be 0.84, the Cronbach alpha reliability coefficient of the Turkish version was found to be 0.83.
Laughter Yoga Satisfaction | four weeks later
  Laughter Yoga Satisfaction Scale: In the first stage of the research, the scale developed by the researcher and the validity-reliability study will be used.
Life Findings Record Form | up to 4 weeks
  The researcher will measure the patient's blood pressure, oxygen saturation, pulse and respiratory rate, body temperature 10 minutes before and 10 minutes after the laughter yoga session and record them on this form.

CONTACTS AND LOCATIONS:
Overall Officials: NURAN TOSUN, PROF., Study Director
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
the study can be shared after publication